CLINICAL TRIAL: NCT06400212
Title: CytoHealth - A Pilot Study of the Phenotypes of the Inflammatory Response to Maximal Exercise.
Brief Title: CytoHealth - A Study of the Inflammatory Response to Exercise
Acronym: CytoHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: York St John University (Other); University of York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 332548Y
Record Dates: First submitted 2024-04-17; First posted 2024-05-06 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Inflammatory Response; Immune System
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Cardiopulmonary Exercise Testing
  Interventions: Other: Cardiopulmonary exercise test

INTERVENTIONS:
Other: Cardiopulmonary exercise test — Participants undergo a cardiopulmonary exercise test following a standardised protocol used in national guidelines

SUMMARY:
By measuring cytokines and chemokines in healthy volunteers of a range of ages and physical fitness, the researchers want to establish how the body's immune system responds to undergoing a single, short test of maximal effort exercise. There is limited research looking at fitness testing and the immune system, particularly in less fit individuals and women. This may not only reveal more about how people respond to the stress of very hard exercise, but it has strong relevance to patients who are undergoing major cancer operations. The researchers know that better fitness improves the patients chances of doing well after a cancer operation, and so patients undergo an exercise test to assess their fitness before a cancer operation. The researchers use this information to guide their treatment during and after their operation. What the researchers do not know is how the immune system responds to the exercise test and how this might be reflected in how they do after the operation.

By undertaking this study, in healthy volunteers, the researchers will not only gain an understanding of how best to assess the immune system during exercise testing, and the logistics of doing this, but it will provide us data that the researchers can compare to cancer patients collected in separate, future study. The potential implication being that information about the immune system could be assessed during exercise testing and enhance how the researchers manage those individuals during and after an operation, potentially improving their outcomes.

To provide a good representation of the general adult population, the researchers will recruit volunteers from two universities and staff at a hospital. Individuals invited to participate will have a blood test to assess their levels of cytokines and chemokines before and after they complete an exercise test. The exercise test will be delivered at one site only, which is a university laboratory.

DETAILED DESCRIPTION:
Using blood tests, the researchers can look at different markers of inflammation circulating in the body. These markers are called cytokines and chemokines. There are many different types of cytokines and chemokines, some of which have been shown to be elevated or lowered in certain medical conditions. A number of them have been shown in studies to be elevated when the body is under stress. One way in which the body can be stressed is through strenuous exercise. The researchers want to understand what happens to cytokine and chemokine release when the participants undertake strenuous exercise in a controlled environment, and in particular the researchers want to measure how the lungs and cardiovascular system are performing and relate that to the markers in the participants blood. By measuring these together, the researchers can better understand how the body's inflammation may be affected by stress and physical fitness.

Ultimately, this information can then be used to inform research looking at patients undergoing surgery. Having a big operation is known to stress the body and the researchers know how well people do after these operations is related to how effectively their lungs and cardiovascular system work prior to the operation (how physically fit they are). What is not clear is what happens to cytokines and chemokines during and after a big operation. The researchers think that higher levels of these markers may be present if someone has lower levels of fitness, and that this would also result in them not doing as well after the operation, but the researchers do not have any studies linking this all together. CytoHealth is a key component of answering this big question as it will provide data on healthy people which the researchers can then use to guide research on patients undergoing surgery.

This study involves recruiting 40 volunteers from the general population from a range of age groups, between aged 18 and 60. In this 40 people the researchers need 20 males and 20 females. In each of these groups of 20 the researchers need 10 to be physically active and 10 to be less physically active. The reason for this categorisation is because existing research in this area is done almost solely in physically active men, and the researchers want our study to be more representative of the general population. Each participant will have to undergo a blood test before and after they exercise to measure their cytokines and chemokines. The exercise will involve a number of monitoring devices to assess how the participant's heart and lungs are functioning during the exercise. Participants involvement in the study concludes once the blood test after exercise is taken. The blood tests taken will go to a specialist laboratory where they will be processed, and the levels variety of cytokines and chemokines will be looked at. This study is a pilot study as there is very limited existing data in this area. This means the researchers are not specifically assessing one particular thing and testing if works or not. Rather the researchers are looking at general trends in the data to provide a basis for further research and importantly, seeing if doing this type of research provides us with scientifically useful information.

The process for the research participant will start with recruitment, which will be done through email communication and posters distributed to staff and students at two universities as well as staff at a large NHS hospital. Individuals who are interested in volunteering will be asked to complete a screening questionnaire which asks their age, sex, physical fitness level and some basic questions about their health. The information from this screening questionnaire can be used to identify the right number people from the groups described above. This questionnaire also outlines what the study involves. Those who are eligible will then be asked to book a slot at the exercise laboratory to attend and take part in the study. They will also be sent a full participant information booklet that will detail what exactly happens in the study.

Once a participant attends on the day they will have to go through a health questionnaire to check they are definitely eligible. They will then go through the study information again with a researcher and if they are happy to proceed, they will be asked to sign a consent form. Once they have consented they are then officially included within the study. At this point they will be allocated a participant identification number (PIN) which will be linked to their identity on a secure spreadsheet which is separate from all data collection. From this point onwards in the study, their data will only be linked to the PIN.

The weight and height of the participant will be recorded, and they will have a blood test taken from their arm. Once this is done they will be asked to sit on the stationary bike. This where they will be connected to an electrocardiogram, a blood pressure cuff, an oxygen saturation probe, a face mask and a finger probe that measures how well the heart is beating, known as a ClearSight finger probe. The face mask is standard monitor used in exercise testing that measures how much oxygen and carbon dioxide is going in and out of the lungs. The participant will then be asked to start pedalling on the bike, which at this point will not be giving any resistance. After a few minutes, a standard programme of increasing resistance is started, such that the participant has to work harder and harder. The aim is to get them to work as hard as they possibly can within about 10 minutes. It is vitally important that the participant does reach the point of exhaustion, or very close to it. Once they reach this point the bike resistance will reduce back down to nothing and the participant will have a few minutes pedalling like this to 'cool down'. They will then be disconnected from the monitoring and a second blood test will be taken.

Once this blood test is done, the participant will be checked to ensure they have appropriately recovered from the exercise and are safe to leave the study. All participants will be given an online shopping voucher worth £50 to compensate them for their time, travel costs and for participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Any individual between the ages of 18 and 60 who has appropriately consented to take part in the study and who does not fulfil any of the 10 exclusion criteria.

Exclusion Criteria:

1. Individuals aged less than 18 years or over 60 years.
2. Individuals who refuse or are unable to give informed consent
3. Individuals with an impairment, injury or disability that prevents them from pedalling on a static bicycle.
4. Individuals who are deemed by a clinician to be classified on the American Society of Anesthesiologists Physical Status Classification System (ASA) as ASA III or ASA IV.
5. Individuals who have had an acute infective or inflammatory illness in the last 7 days.
6. Individuals who have undertaken moderate or high intensity exercise in the 24 hours prior to the exercise testing.
7. Individuals who have a cardiac or respiratory condition which poses significant restrictions on their exercise capacity, as assessed by a clinician. Including but not limited to the following: recent myocardial infarction, acquired or inherited arrythmias or cardiomyopathies, presence of an implantable defibrillator or pacemaker, uncontrolled or severe COPD, uncontrolled asthma, pulmonary hypertension, pulmonary fibrosis.
8. Individuals who are pregnant.
9. Individuals who are known to have an active malignancy or have undergone treatment for cancer in the last year.
10. Individuals who are currently an inpatient in a hospital.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Serum cytokines | Sample taken immediately prior and immediately after exercise testing
  Pre-designed multiplex flow assay panels (LEGENDplexTM BioLegend, San Diego, CA, USA) for detections of cytokines and chemokines will be used. These will be a human cytokines panel (IL- 1,2, 4, 5, 6, 9, 10, 13, 17A, 17F, 21 and 22. IFNg and TNFa) to evaluate the presence of systemic cytokine expression, and a proinflammatory chemokines panel [MCP-1 (CCL2), RANTES (CCL5), IP-10 (CXCL10), Eotaxin (CCL11), TARC (CCL17), MIP-1α (CCL3), MIP-1β (CCL4), MIG (CXCL9), MIP-3α (CCL20), ENA-78 (CXCL5), GROα (CXCL1), I-TAC (CXCL11) and IL-8 (CXCL8)] for the assessment of chemokine profiles. Serum levels of cytokines and chemokines will be determined from flow cytometry results using the free manufacturer data analysis software (www.biolegend.com/legendplex) and will be expressed as concentrations (pg/ml) calculated from a calibration curve

SECONDARY OUTCOMES:
VO2 (oxygen consumption of participant during exercise) | Data measured continuously during exercise testing (average duration of exercise test is 20 minutes)
  Measured in ml/kg/min using gas analysis which is connected to participant via a face mask
VCO2 (carbon dioxide exhaled by participant during exercise) | Data measured continuously during exercise testing (average duration of exercise test is 20 minutes)
  Measured in ml/kg/min using gas analysis which is connected to participant via a face mask
Heart rate including maximum heart rate | Data measured continuously during exercise testing (average duration of exercise test is 20 minutes)
  Measured using electrocardiogram in beats per minute (BPM)
Respiratory exchange ratio (volume of expired carbon dioxide compared to volume of oxygen consumed) including the peak RER | Data measured continuously during exercise testing (average duration of exercise test is 20 minutes)
  No units as ratio.
Anaerobic threshold | Data measured continuously during exercise testing (average duration of exercise test is 20 minutes)
  Determined by the v-slope method of graphically comparing VO2 with VCO2 with the units being ml/kg/min
Stroke volume | Data taken during exercise testing at 20 second intervals (average duration of exercise test is 20 minutes)
  Determined by ClearSight finger cuff monitor with the unit mls
Borg rate of perceived exertion (RPE) | Immediately at end of exercise test
  Participant asked to rate level of exertion at end of test using rate of perceived exertion scale (1-10).

CONTACTS AND LOCATIONS:
Overall Officials: John O'Rourke, Principal Investigator — Academic Clinical Fellow
Locations (1):
- York and Scarborough Teaching Hospitals NHS Foundation Trust, York, North Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No